CLINICAL TRIAL: NCT04796740
Title: Postoperative Arterial or Venous Thrombembolism After Robot- Assisted Surgery in Major Urological Procedures is in Some Cases a Severe Complication.
Brief Title: Thrombembolism After Robot- Assisted Surgery in Urology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, Clinical Professor, University Hospital Schleswig-Holstein
Other Study IDs: IN-UDV_01
Record Dates: First submitted 2020-12-17; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Urologic Cancer; Thrombosis; Embolism; Surgery--Complications
Keywords: thrombembolism after robot-assisted surgery
MeSH Terms: conditions — Urologic Neoplasms; Thrombosis; Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Cancer patients have an increased risk of perioperative complications undergoing surgery procedures. Postoperative complications caused by thrombembolic events after robot- assisted surgery in major urological procedures have been reported and associated with an increased lenght of stay in the hospital. We therefore aimed to investigate in a retrospective analysis 250 patients undergoing robotic-assisted radical cystectomy and prostatectomy procedures for risk factors for thrombembolic events in this specific patient population.

DETAILED DESCRIPTION:
Postoperative arterial or venous thrombembolism after robotic- assisted surgery in major urological procedures are reported severe complications in this patient population.

After having studied the available literature on this particular topic the investigators have decided to prepare a retrospective analysis of approximately 250 robot- assisted radical cystectomy and radical prostatectomy surgical procedures. In due consideration of perioperative prophylaxis of thrombembolic Events we determine the clinical and radiological signs of venous or arterial thrombembolism postoperatively with a particular focus on early postoperative pulmonary embolism events.

This is a retrospective analysis of 250 robotic-assisted radical cystectomy and radical prostatectomy surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* scheduled for urological surgery (cystectomy and/or prostatectomy)
* signed basical declaration of consent

Exclusion Criteria:

* absent or unsigned basical declaration of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collective of patients with bladder- and/or prostate cancer scheduled for laporoscopic robot-assited radical cystectomy and/or prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative thrombembolism | through study completion, an average of 1 year
  Arterial and venous thrombembolism after surgery

SECONDARY OUTCOMES:
acute renal failure | through study completion, an average of 1 year
  acute renal failure
pulmonary oedema | through study completion, an average of 1 year
  pulmonary oedema
pneumonia | through study completion, an average of 1 year
  pneumonia
wound infection | through study completion, an average of 1 year
  wound infection
Major adverse cardiovascular events (MACE) | through study completion, an average of 1 year
  nonfatal stroke, nonfatal myocardial infarction and cardiovascular death
ocular complications | through study completion, an average of 1 year
  ocular complications
delirium | through study completion, an average of 1 year
  delirium

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, Prof. Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abel EJ, Wong K, Sado M, Leverson GE, Patel SR, Downs TM, Jarrard DF. Surgical operative time increases the risk of deep venous thrombosis and pulmonary embolism in robotic prostatectomy. JSLS. 2014 Apr-Jun;18(2):282-7. doi: 10.4293/108680813X13693422518551. PMID 24960494
- [Background] Mehrazin R, Piotrowski Z, Egleston B, Parker D, Tomaszweski JJ, Smaldone MC, Abbosh PH, Ito T, Bloch P, Iffrig K, Bilusic M, Chen DY, Viterbo R, Greenberg RE, Uzzo RG, Kutikov A. Is extended pharmacologic venous thromboembolism prophylaxis uniformly safe after radical cystectomy? Urology. 2014 Nov;84(5):1152-6. doi: 10.1016/j.urology.2014.06.058. Epub 2014 Oct 24. PMID 25443917
- [Background] Tyritzis SI, Wallerstedt A, Steineck G, Nyberg T, Hugosson J, Bjartell A, Wilderang U, Thorsteinsdottir T, Carlsson S, Stranne J, Haglind E, Wiklund NP; LAPPRO Steering Committee. Thromboembolic complications in 3,544 patients undergoing radical prostatectomy with or without lymph node dissection. J Urol. 2015 Jan;193(1):117-25. doi: 10.1016/j.juro.2014.08.091. Epub 2014 Aug 23. PMID 25158271
- [Background] Hope WW, Demeter BL, Newcomb WL, Schmelzer TM, Schiffern LM, Heniford BT, Sing RF. Postoperative pulmonary embolism: timing, diagnosis, treatment, and outcomes. Am J Surg. 2007 Dec;194(6):814-8; discussion 818-9. doi: 10.1016/j.amjsurg.2007.08.014. PMID 18005777